CLINICAL TRIAL: NCT00006325
Title: Safety, Tolerability, Antiviral Activity, and Pharmacokinetics of PEG-Intron in HIV-1 Infected Children
Brief Title: Safety, Tolerability, and Anti-HIV Activity of PEG-Intron in HIV-Positive Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P1017; PACTG P1017; ACTG P1017; 11652 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2000-10-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Polyethylene Glycols; Interferon Alfa-2b; HIV-1; Dose-Response Relationship, Drug; Drug Therapy, Combination; Virus Inhibitors; Anti-HIV Agents; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — peginterferon alfa-2b

INTERVENTIONS:
Drug: Peginterferon alfa-2b

SUMMARY:
The purpose of this study is to see if PEG-Intron is safe and tolerated when given to children, to see how much gets into the blood and how long it stays in the blood, and to see how well it works to reduce viral load (level of HIV in the blood).

PEG-Intron is an experimental drug that works differently than other anti-HIV medications. It decreases the ability of HIV to infect the T cells (a special type of cell that helps fight infection). PEG-Intron has been approved by the Food and Drug Administration (FDA) to treat hepatitis C in adults, but in this study, it is being used as an investigational agent for the treatment of HIV/AIDS. It has not been tested in children before and experience with PEG-Intron in adults is limited. (This protocol has been changed to reflect FDA approval of PEG-Intron for treating hepatitic C in adults.)

DETAILED DESCRIPTION:
The current optimal clinical management of HIV infection involves therapy with combinations of nucleoside and nonnucleoside reverse transcriptase inhibitors and HIV protease inhibitors. These regimens, though effective, do not completely eliminate HIV and the development of drug resistance is a major clinical problem. Interferons have been proposed as a possible treatment of HIV. Interferon-alfa inhibits HIV replication in vitro, and HIV-infected patients appear to have reduced production of interferons. Previous short-term clinical studies in adults showed anti-HIV activity, although there were safety and tolerability problems associated with the higher dose regimens used. This study will utilize a rising multiple-dose design to assess the safety, tolerability, and pharmacokinetics of single and multiple doses of PEG-Intron in HIV-infected children.

In a dose-escalation study, patients add weekly PEG-Intron to their antiretroviral therapy for up to 6 weeks. The first 2 doses are received in the clinic where parents/guardians are trained to administer injections, and succeeding doses are given at home.

Patients are enrolled from 2 cohorts. An older cohort of ages 2 to 16 years receives PEG-Intron at the lowest drug level. If the dose is tolerated, patients are added and if safety criteria are met, patients are enrolled in the next higher dose level. The dose level will be increased similarly for up to 4 doses. An optimal dose level is chosen.

Cohort II patients are a younger group ranging from 3 months to under 2 years of age. Patients initially receive the next lower PEG-Intron dose to the optimal dose identified in Cohort I [AS PER AMENDMENT 07/23/01: or 1 microg/kg if the optimal dose proves to be 1 microg/kg]. If this dose is safely tolerated, additional patients are added. If this dose level meets safety criteria, patients are enrolled to receive the optimal dose level. Patients are evaluated with the same safety criteria as Cohort I. Patients in both cohorts who have at least a 0.5 log reduction in HIV RNA at 28 days of treatment are offered continued treatment for a total of 60 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-infected infants and children aged 3 months to 16 years.
* Have been on stable anti-HIV drugs for at least 16 weeks if over 6 months of age. Infants aged 3 to 6 months must be on stable anti-HIV drugs for at least 6 weeks. Children should be receiving at least 3 anti-HIV drugs.
* Have a viral load of more than 5,000 copies/ml.
* Have written informed consent from parent or guardian and, if able, can give written consent themselves.
* Are able to follow the schedule in the protocol.
* Have a parent/guardian who is willing to comply with study requirements.
* (This study has been changed to allow any combination of 3 anti-HIV drugs and to remove CD4 requirements.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are breast-feeding or pregnant or not using birth control, if a female.
* Have abnormal thyroid activity.
* Have severe HIV symptoms.
* Have opportunistic (AIDS-related) infections or history of such infections within the preceding 2 months.
* Have participated in a clinical trial of an experimental drug in the previous month.
* Have a positive test result for hepatitis B or C.
* Have an allergy to E. coli.
* Have a mental disorder.
* Have a history of drug dependence and measure positive when screened.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Luzuriaga, Study Chair; Andrea Kovacs, Study Chair
Locations (15):
- United States (15):
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Schneider Children's Hosp, New Hyde Park, New York
  - Harlem Hosp Ctr, New York, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Texas Children's Hosp / Baylor Univ, Houston, Texas